CLINICAL TRIAL: NCT02782715
Title: Real-time MRI-Guided Stereotactic Body Radiation Therapy and Microwave Ablation for Non-Operable Renal Cell Carcinoma
Brief Title: Microwave Ablation With MRI-Guided SBRT Boost in Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW15103; 2016-0286 (Other: Institutional Review Board); NCI-2016-00775 (Registry Identifier: NCI Trial ID); A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison); Protocol Version 4/16/2019 (Other: UW Madison)
Record Dates: First submitted 2016-05-19; First posted 2016-05-25 (Estimated); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiotherapy & Microwave Ablation (Experimental): 3+3 dose-escalation wherein three dose levels of stereotactic body radiation therapy (SBRT) would be evaluated:
  1. Dose level I: 6 Gy x 5 fractions
  2. Dose level II: 8 Gy x 5 fractions
  3. Dose level III: 10 Gy x 5 fractions
  Radiation treatments will be delivered two to three times a week, with five fractions completed over two weeks.
  Four to six weeks after radiation treatment, patients will undergo repeat CT or MRI imaging to assess tumor response and suitability for microwave ablations.
  Eight weeks after the conclusion of SBRT, patients will undergo microwave ablation (approximately 12 weeks after registration).
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Microwave Ablation (MWA)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients will be treated on study with a course of SBRT treatment by a radiation oncologist. Three SBRT dose levels targeting the primary tumor will be evaluated; level I: 6 Gy x 5 fractions (a common palliative dose), level II: 8 Gy x 5 fractions, and level III: 10 Gy x 5 fractions (a common definitive dose).
Procedure: Microwave Ablation (MWA) — Performed under sedation using ultrasound and computed tomography (CT) guidance for percutaneous antenna placement and confirmation. Depending on size and location of tumor, one to three antennas (Certus 140; NeuWave Medical) will be used. The system is an FDA-approved, high-powered third-generation MW device that uses CO2 gas cooling to prevent shaft heating. The gas cooling allows the probes to be stuck into tissue by creating a small ice ball at the tip using the Joule-Thomson method, similar to the tissue cooling mechanism of cryoablation systems. Probes are 17-gauge, and various ablation zone configurations are available depending on the probe selected. An ablation protocol using the 65W power setting for 5 minutes will be used for most patients. Ultrasound will be used for real-time monitoring of the extent of ablation to achieve a 5mm margin beyond tumor, and immediate post-procedure imaging performed using contrast-enhanced CT (CECT) for patients with adequate renal functions.

SUMMARY:
The specific aims of this study are:

1. To determine the safety and feasibility of treating patients with a combination of MRI guided stereotactic body radiation therapy and microwave ablation.
2. To assess short and long-term toxicity rates of patients treated with a combined modality approach.
3. To assess local control, survival, and pathologic response to treatment

DETAILED DESCRIPTION:
Renal cell carcinoma is traditionally managed via a surgical approach. Increasingly, local therapy with radiofrequency and microwave ablation is being utilized as an alternative for patients who may not tolerate a nephrectomy or who refuse one. Although local control rates for small lesions are excellent, they drop off precipitously for lesions over 4 cm. Furthermore, lesions in critical areas such as the renal hilum may be difficult to treat with this method. Stereotactic body radiation therapy (SBRT) has had a long record of treating patients with inoperable tumors in locations such as the lung and central nervous system, and there is increasing evidence that it may be useful for patients with renal cell carcinoma. The recent emergence of MRI-guided radiation therapy allows for direct visualization of tumors during treatment, and may potentially allow clinicians to treat tumors more precisely. This phase I study will treat renal cell carcinoma patients using a combination of MRI-guided stereotactic body radiation therapy and microwave ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with imaging findings consistent with renal cell carcinoma
* Deemed medically inoperable per urology evaluation
* Tumor size >4cm in largest dimension
* ECOG performance status of <2
* Signed informed consent document(s)
* Patients with metastatic disease will not be excluded

Exclusion Criteria:

* Patients who fail MRI screening
* Pregnant or nursing women
* History of prior radiation therapy to the upper abdomen
* History of invasive cancer in the last 3 years (except for appropriately treated low-rist prostate cancer, treated non-melanoma/melanoma skin cancer, appropriately treated ductal carcinoma in situ or early stage invasive carcinoma of breast and appropriately treated in-situ/early stage cervical/endometrial cancer)
* Treatment with a non-approved or investigational drug within 28 days of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bassetti, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from June 2018 to September 2022.
Period: Overall Study
Arm/Group | Radiotherapy & Microwave Ablation
Started | 3
On Treatment | 3
Off Treatment | 3
Completed Ablation | 2
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiotherapy & Microwave Ablation
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  70-79 years old | 2
  80-89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity With SBRT Combined With Microwave Ablation for Renal Cell Carcinoma
Description: Dose-limiting toxicity (DLT) will be defined as grade 4 or higher non-hematologic toxicity attributable to treatment. This will exclude toxicities not caused by treatment, such as pain due to tumor progression. Toxicities will be defined per NCI CTCAE v5.0.
Time Frame: Until 30 days after ablation (up to 12 weeks on study)
Population: 1 participant did not undergo ablation
Measure: Number; unit: dose limiting toxicities
Arm/Group | Radiotherapy & Microwave Ablation
Number analyzed (Participants) | 2
dose limiting toxicities | 0

2. Secondary Outcome: Local Control Rate Per RECIST Criteria as Reported by Count of Participants
Description: Radiologic response per RECIST criteria and volumetric measurements.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy & Microwave Ablation
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Progression Free Survival
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy & Microwave Ablation
Number analyzed (Participants) | 2
Participants | 2

4. Secondary Outcome: Overall Survival
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy & Microwave Ablation
Number analyzed (Participants) | 2
Participants | 2

5. Secondary Outcome: Tumor Pathology of Post-SBRT Specimen (H&E Staining)
Description: H&E staining for percentage of viable tumor remaining as measured by the presence of necrosis, fibrosis, hyalinization, and/or calcification, compared to pre-SBRT pathology
Time Frame: 8 weeks
Population: tumor pathology was not analyzed as study was terminated early, no data collected
Arm/Group | Radiotherapy & Microwave Ablation
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Tumor Pathology of Post-SBRT Specimen (Pathologic Evaluation)
Description: Pathologic evaluation for percentage of viable tumor remaining as measured by the presence of necrosis, fibrosis, hyalinization, and/or calcification, compared to pre-SBRT pathology
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Arm/Group | Radiotherapy & Microwave Ablation
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy & Microwave Ablation (N=3)
anemia (Blood and lymphatic system disorders) | 1
lymphopenia (Immune system disorders) | 1
headache (General disorders) | 1
Fatigue (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT02782715/Prot_SAP_000.pdf